CLINICAL TRIAL: NCT06250088
Title: Efficacy of Enamel Matrix Derivatives Adjunctive to Closed-apex Teeth Autotransplantation A Randomized Clinical Trial
Brief Title: Emdogain Adjunctive to Autotransplantation
Acronym: ATTEMD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Ignacio Pedrinaci Peñalver, Principal investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATT_EMD_RCT
Record Dates: First submitted 2024-01-23; First posted 2024-02-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Autotransplantation; Emdogain; Autologous Transplantation; Enamel Matrix Derivatives
Keywords: Emdogain and tooth autotransplantation
MeSH Terms: interventions — enamel matrix proteins; emerin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emdogain (EMD) (Active Comparator)
  Interventions: Biological: Emdogain (EMD) - test; Procedure: Sham group
- Control (Sham Comparator)
  Interventions: Procedure: Sham group

INTERVENTIONS:
Biological: Emdogain (EMD) - test — Initially, tooth sectioning of the hopeless tooth (receptor) will be carried out using fissure carbide burs, and the resulting fragments will be extracted with a minimally invasive approach. A multiple drilling axis tooth-supported surgical guide will be used to prepare the recipient site in accordance with the 3D planning. Additional alveoloplasty procedures will be performed with round diamond burs if necessary to adapt the computer assisted rapid prototyping (CARP) model to the virtual planning position. The donor tooth will be extracted as atraumatically as possible, utilizing a piezoelectric if ostectomy is required, and avoiding the use of elevators or forceps over the root surface. Extraorally, (Emdogain) EMD will be applied to the root surface of the donor tooth. Sutures will be applied to closely adapt the soft tissues around the autotransplanted tooth. A semi-rigid orthodontic wire will be used to splint the tooth to the mesial and distal adjacent teeth
  Arms: Emdogain (EMD)
Procedure: Sham group — Initially, tooth sectioning of the hopeless tooth (receptor) will be carried out using fissure carbide burs, and the resulting two fragments will be extracted with a minimally invasive approach. A multiple drilling axis tooth-supported surgical guide will be used to prepare the recipient site in accordance with the 3D planning. Additional alveoloplasty procedures will be performed with round diamond burs if necessary to adapt thecomputer assisted rapid prototyping (CARP) model to the virtual planning position. The donor tooth will be extracted as atraumatically as possible, utilizing a piezoelectric surgical instrument if ostectomy is required, and avoiding the use of elevators or forceps over the root surface. No Emdodain (EMD). Sutures will be applied to closely adapt the soft tissues around the autotransplanted tooth. A semi-rigid orthodontic wire will be used to splint the tooth to the mesial and distal adjacent teeth

SUMMARY:
The goal of this randomized clinical trial is to compare the adjunctive use of enamel matrix derivatives in the treatment of tooth autotransplantation in terms of clinical attachment level. The main question it aims to answer. What is the benefit, in terms of clinical attachment level and probing depths, of using enamel matrix derivatives adjunctive to tooth autotransplantation? Participants will be subjected to a digitally guided surgery of tooth autotransplantation. The protocol of the test group will be supplemented with the application of enamel matrix derivatives before the placement of the transplanted tooth into the surgically produced alveolus.

ELIGIBILITY:
Inclusion Criteria: Adult patients attending the University Complutense of Madrid for dental treatment were eligible to participate in the study if they met the following criteria:

* adults (≥18 years old) capable of providing informed consent, teeth deemed-unrestorable in need of replacement
* presence of a viable, healthy, periodontally stable, and nonfunctional tooth (e.g., third molar) suitable for autotransplantation
* periodontally healthy individuals or those with stable periodontal conditions after periodontal therapy.

Exclusion Criteria:

* clinical attachment loss of the donor teeth (CAL less 6 mm)
* compromised general health or patients with systemic diseases that could influence the therapy outcome (uncontrolled diabetes mellitus, bone disorders, etc.)
* pregnant or nursing women
* chronic use of corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or immune-modulator drugs
* patients requiring medications that affect bone metabolism (bisphosphonates
* chronic oral mucosa diseases
* evident signs of severe bruxism or clenching habits
* smokers of more than 10 cigarettes per day
* non-compliant patients with 25% plaque index at the time of re-evaluation after non-surgical periodontal therapy and oral hygiene instructions
* patients unable to attend study-related procedures and follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | through study completion, an average of 1 year
  measured as the distance in mm from the CEJ to the bottom of the pocket will be the primary outcome of this study.

SECONDARY OUTCOMES:
Radiographic bone level | through study completion, an average of 1 year
  Changes in marginal bone levels (MBLs), measured as the change in interproximal bone levels between 4 weeks after autotransplantation, six months and one year postoperatively. MBLs are defined as the distance between the cementoenamel junction (CEJ) and to the crestal bone level at the mesial and distal aspect . These measurements will also be recorded at the adjacent teeth/implants. For standardization of the radiographic technique, a customized bite block will be constructed for each patient using a parallel technique X-ray film holder (i.e.Rinn System, x-ray system or similar) and heavy silicone. The obtained digital radiographs will be evaluated using the image software (OsiriX Imaging Software, Geneva, Switzerland), with previous calibration of the images by inserting a small metal object of known measures in the bite block
Digital image assessment. Position of the Alveolar Ridge Measurements | at the study completion. an average of 1 year
  For each patient, the baseline and the last follow-up visit STL files and Digital Imaging and Communications in Medicine (DICOM) files will be superimposed for best-fit alignment. Alveolar ridge width changes will also be evaluated at the buccal and lingual mesial, mid, and distal sites. A sagittal section at each area of interest will be made. Horizontal alveolar ridge width linear changes will be quantified in mm at three predetermined reference points established at 1, 3, and 5mm from the baseline gingival margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No